CLINICAL TRIAL: NCT00972283
Title: NN1250-3582: A 52-week Randomised, Controlled, Open Label, Multicentre, Multinational Treat-to-target Trial Comparing Efficacy and Safety of SIBA and Insulin Glargine Both Administered Once Daily in a Basal-bolus Regimen With Insulin Aspart as Mealtime Insulin ± Treatment With Metformin, ± Pioglitazone in Subjects With Type 2 Diabetes Currently Treated With Insulin Qualifying for Intensified Treatment/NN1250-3667: An Extension Trial to NN1250-3582 Comparing Safety and Efficacy of NN1250 and Insulin Glargine, Both With Insulin Aspart as Meal-time Insulin ± OADs in Type 2 Diabetes (BEGIN™: BB)
Brief Title: Comparison of NN1250 With Insulin Glargine Plus Insulin Aspart With/Without Metformin and With/Without Pioglitazone in Type 2 Diabetes
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3582; 2008-005777-35 (EudraCT Number); U1111-1111-8648 (Other: WHO); 2009-015816-17 (EudraCT Number); U1111-1114-9067 (Other: WHO); NCT01193322 (obsolete NCT alias)
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2015-11-13 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg OD (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- IGlar OD (Active Comparator)
  Interventions: Drug: insulin glargine; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec — Injected subcutaneously (under the skin) with main evening meal. Dose was individually adjusted.
  Arms: IDeg OD
Drug: insulin glargine — Injected subcutanoeusly (under the skin) according to approved label. Dose was individually adjusted.
  Arms: IGlar OD
Drug: insulin aspart — Injected subcutaneously (under the skin) at each main meal. Dose was individually adjusted.

SUMMARY:
This trial is conducted in Africa, Asia, Europe, and the United States of America (USA).

The aim of this clinical trial is to compare NN1250 (insulin degludec (IDeg)) with insulin glargine (IGlar) plus insulin aspart (IAsp) with/without metformin and with/without pioglitazone in subjects with type 2 diabetes (main period) followed by investigating the long-term safety in terms of comparing NN1250 with insulin glargine plus insulin aspart with or without metformin and with or without pioglitazone in subjects with type 2 diabetes.

All oral anti-diabetic drug (OAD) treatment will be discontinued, if applicable, when trial participant enters the trial (NN1250-3582) with the exception of metformin and pioglitazone.

Subjects who consent to participate in the extension trial (NN1250-3667) will continue to receive the treatment to which they were randomly allocated in the 52 week trial NN1250-3582.

The main period is registered internally at Novo Nordisk as NN1250-3582 while the extension period is registered as NN1250-3667.

ELIGIBILITY:
Inclusion Criteria:

* For MAIN period (NN1250-3582):
* Type 2 diabetes mellitus for at least 6 months
* Ongoing daily treatment with insulin (premix, self-mix, basal only, basal bolus) for at least 3 months with/without oral anti-diabetics drug (OAD) prior to trial start
* HbA1c 7.0-10.0 % (both inclusive)
* Body Mass Index (BMI) below or equal to 40.0 kg/m^2
* For EXTENSION period (NN1250-3667):
* Completion of the 52 week treatment period in NN1250-3582

Exclusion Criteria:

* For MAIN period (NN1250-3582):
* Treatment with other insulin regimens than premix, self-mix, basal only, basal bolus within 3 months
* Cardiovascular disease within the last 6 months
* Uncontrolled treated/untreated severe hypertension
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures
* Cancer and medical history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1006 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2010-10-28 (Actual); Study Completion 2010-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (123):
- United States (64):
  - Novo Nordisk Investigational Site, Alexander City, Alabama
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Goodyear, Arizona
  - Novo Nordisk Investigational Site, Peoria, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, Los Gatos, California
  - Novo Nordisk Investigational Site, Salinas, California
  - Novo Nordisk Investigational Site, Santa Monica, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Milford, Connecticut
  - Novo Nordisk Investigational Site, Norwalk, Connecticut
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Gainesville, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Lake Mary, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Fort Valley, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Nampa, Idaho
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, New Albany, Indiana
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, North East, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Eagan, Minnesota
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Lincoln, Nebraska
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Danville, Pennsylvania
  - Novo Nordisk Investigational Site, Kingston, Pennsylvania
  - Novo Nordisk Investigational Site, Melrose Park, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Wilkes-Barre, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Newberry, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
- Bulgaria (5):
  - Novo Nordisk Investigational Site, Dimitrovgrad
  - Novo Nordisk Investigational Site, Rousse
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Stara Zagora
  - Novo Nordisk Investigational Site, Varna
- Germany (8):
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Wangen
  - Novo Nordisk Investigational Site, Warburg
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- Novo Nordisk Investigational Site, Dublin, Ireland
- Italy (13):
  - Novo Nordisk Investigational Site, Bari
  - Novo Nordisk Investigational Site, Bergamo
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Chieti Scalo
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Foggia
  - Novo Nordisk Investigational Site, Gazi
  - Novo Nordisk Investigational Site, Messina
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Perugia
  - Novo Nordisk Investigational Site, Pisa
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Torino
- Romania (5):
  - Novo Nordisk Investigational Site, Baia Mare, Maramureş
  - Novo Nordisk Investigational Site, Suceava, Suceava
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Constanța
  - Novo Nordisk Investigational Site, Timișoara
- Russia (7):
  - Novo Nordisk Investigational Site, Arkhangelsk
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Krasnoyarsk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Perm
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Yaroslavl
- Slovakia (2):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Lučenec
- South Africa (3):
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Bloemfontein
- Spain (11):
  - Novo Nordisk Investigational Site, A Coruña
  - Novo Nordisk Investigational Site, Alcorcón
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, L'Hospitalet de Llobregat
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Mostoles - Madrid -
  - Novo Nordisk Investigational Site, Sabadell
  - Novo Nordisk Investigational Site, San Juan
  - Novo Nordisk Investigational Site, Valencia
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Mersin

REFERENCES:
- [Result] Ratner RE, Gough SC, Mathieu C, Del Prato S, Bode B, Mersebach H, Endahl L, Zinman B. Hypoglycaemia risk with insulin degludec compared with insulin glargine in type 2 and type 1 diabetes: a pre-planned meta-analysis of phase 3 trials. Diabetes Obes Metab. 2013 Feb;15(2):175-84. doi: 10.1111/dom.12032. Epub 2012 Dec 3. PMID 23130654
- [Result] Heller S, Mathieu C, Kapur R, Wolden ML, Zinman B. A meta-analysis of rate ratios for nocturnal confirmed hypoglycaemia with insulin degludec vs. insulin glargine using different definitions for hypoglycaemia. Diabet Med. 2016 Apr;33(4):478-87. doi: 10.1111/dme.13002. Epub 2015 Dec 13. PMID 26484727
- [Result] Sorli C, Warren M, Oyer D, Mersebach H, Johansen T, Gough SC. Elderly patients with diabetes experience a lower rate of nocturnal hypoglycaemia with insulin degludec than with insulin glargine: a meta-analysis of phase IIIa trials. Drugs Aging. 2013 Dec;30(12):1009-18. doi: 10.1007/s40266-013-0128-2. PMID 24170235
- [Result] Einhorn D, Handelsman Y, Bode BW, Endahl LA, Mersebach H, King AB. PATIENTS ACHIEVING GOOD GLYCEMIC CONTROL (HBA1c <7%) EXPERIENCE A LOWER RATE OF HYPOGLYCEMIA WITH INSULIN DEGLUDEC THAN WITH INSULIN GLARGINE: A META-ANALYSIS OF PHASE 3A TRIALS. Endocr Pract. 2015 Aug;21(8):917-26. doi: 10.4158/EP14523.OR. Epub 2015 Jun 29. PMID 26121451
- [Result] Russell-Jones D, Gall MA, Niemeyer M, Diamant M, Del Prato S. Insulin degludec results in lower rates of nocturnal hypoglycaemia and fasting plasma glucose vs. insulin glargine: A meta-analysis of seven clinical trials. Nutr Metab Cardiovasc Dis. 2015 Oct;25(10):898-905. doi: 10.1016/j.numecd.2015.06.005. Epub 2015 Jun 18. PMID 26232910
- [Result] Vora J, Christensen T, Rana A, Bain SC. Insulin degludec versus insulin glargine in type 1 and type 2 diabetes mellitus: a meta-analysis of endpoints in phase 3a trials. Diabetes Ther. 2014 Dec;5(2):435-46. doi: 10.1007/s13300-014-0076-9. Epub 2014 Aug 1. PMID 25081590
- [Result] Aye MM, Atkin SL. Patient safety and minimizing risk with insulin administration - role of insulin degludec. Drug Healthc Patient Saf. 2014 Apr 30;6:55-67. doi: 10.2147/DHPS.S59566. eCollection 2014. PMID 24812526
- [Result] Garber AJ, King AB, Del Prato S, Sreenan S, Balci MK, Munoz-Torres M, Rosenstock J, Endahl LA, Francisco AM, Hollander P; NN1250-3582 (BEGIN BB T2D) Trial Investigators. Insulin degludec, an ultra-longacting basal insulin, versus insulin glargine in basal-bolus treatment with mealtime insulin aspart in type 2 diabetes (BEGIN Basal-Bolus Type 2): a phase 3, randomised, open-label, treat-to-target non-inferiority trial. Lancet. 2012 Apr 21;379(9825):1498-507. doi: 10.1016/S0140-6736(12)60205-0. PMID 22521072
- [Result] Hollander P, King AB, Del Prato S, Sreenan S, Balci MK, Munoz-Torres M, Rosenstock J, Hansen CT, Niemeyer M, Garber AJ. Insulin degludec improves long-term glycaemic control similarly to insulin glargine but with fewer hypoglycaemic episodes in patients with advanced type 2 diabetes on basal-bolus insulin therapy. Diabetes Obes Metab. 2015 Feb;17(2):202-6. doi: 10.1111/dom.12411. Epub 2014 Nov 27. PMID 25387855
- [Result] Freemantle N, Mamdani M, Vilsboll T, Kongso JH, Kvist K, Bain SC. IDegLira Versus Alternative Intensification Strategies in Patients with Type 2 Diabetes Inadequately Controlled on Basal Insulin Therapy. Diabetes Ther. 2015 Dec;6(4):573-591. doi: 10.1007/s13300-015-0142-y. Epub 2015 Nov 18. PMID 26582052
- [Result] Evans M, Chubb B, Gundgaard J. Cost-effectiveness of Insulin Degludec Versus Insulin Glargine in Adults with Type 1 and Type 2 Diabetes Mellitus. Diabetes Ther. 2017 Apr;8(2):275-291. doi: 10.1007/s13300-017-0236-9. Epub 2017 Feb 16. PMID 28210866
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 123 sites in 12 countries: Bulgaria (8 sites), Germany (8), Hong Kong (1), Ireland (4), Italy (11), Romania (5), Russia (6), Slovakia (4), South Africa (5), Spain (9), Turkey (3) and the United States (U.S.) (59). Some sites did not enroll subjects in the extension period. One site from United States was closed.
Pre-assignment Details: All subjects who completed the 52-week main trial (NN1250-3582, NCT00972283) and were found to be eligible for the extension trial were offered to participate in the 26-week extension trial (NN1250-3667). The total duration of treatment was up to 78 weeks (52 weeks + 26 weeks).
Groups:
- IDeg OD: Insulin degludec (IDeg) was given subcutaneously once daily (OD) with main evening meal with insulin aspart (IAsp) as mealtime insulin with or without subject's pre-trial metformin with or without pioglitazone. The regimen was given for a treatment duration of 52 weeks in the main period and for an additional 26 weeks in the extension period.
- IGlar OD: Insulin glargine (IGlar) was given subcutaneously once daily (OD), according to labelling instructions with insulin aspart (IAsp) as mealtime insulin with or without subject's pre-trial metformin with or without pioglitazone. IGlar was given for a treatment duration of 52 weeks in the main period and for an additional 26 weeks in the extension period.
Period: Main: Week 0 to 52 (NN1250-3582)
Arm/Group | IDeg OD | IGlar OD
Started | 755 | 251
Full Analysis Set | 744 (11 subjects were excluded due to closure of a site) | 248 (3 subjects were excluded due to closure of a site)
Exposed | 753 (2 subjects were withdrawn prior to exposure to trial products) | 251
Completed | 618 | 211
Not Completed | 137 | 40
Not completed — Adverse Event | 31 | 9
Not completed — Lack of Efficacy | 3 | 0
Not completed — Protocol Violation | 23 | 12
Not completed — Withdrawal criteria | 8 | 2
Not completed — Unclassified | 72 | 17
Period: Extension: Week 53 to 78 (NN1250-3667)
Arm/Group | IDeg OD | IGlar OD
Started | 566 (52 subjects did not continue into the extension from main trial) | 191 (20 subjects did not continue into the extension from main trial)
Completed | 539 | 183
Not Completed | 27 | 8
Not completed — Adverse Event | 4 | 0
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 5 | 0
Not completed — Withdrawal criteria | 6 | 2
Not completed — Unclassified | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg OD | IGlar OD | Total
Number analyzed (Participants) | 744 | 248 | 992
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.1) | 58.1 (10.0) | 58.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 339 | 115 | 454
  Male | 405 | 133 | 538
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (0.8) | 8.4 (0.9) | 8.3 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Main Trial (Primary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 52 Weeks of Treatment
Description: Change from baseline in HbA1c after 52 weeks of treatment
Time Frame: Week 0, Week 52
Population: Full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 744 | 248
percentage of glycosylated haemoglobin | -1.17 (1.03) | -1.29 (0.98)

2. Secondary Outcome: Extension Trial (Secondary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 78 Weeks of Treatment
Description: Change from baseline in HbA1c after 78 weeks of treatment
Time Frame: Week 0, Week 78
Population: The FAS included all randomised subjects in the main trial including subjects carried through to the extension trial and missing data was imputed using LOCF
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 744 | 248
percentage of glycosylated haemoglobin | -0.95 (1.13) | -1.15 (0.99)

3. Secondary Outcome: Main Trial (Secondary Endpoint): Mean of 9-point Self Measured Plasma Glucose Profile (SMPG) at Week 52
Description: Mean of 9-point SMPG at 52 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime, at 4 am and before breakfast.
Time Frame: Week 52
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. For 36 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 715 | 241
mmol/L | 7.3 (1.8) | 6.9 (1.5)

4. Secondary Outcome: Extension Trial (Secondary Endpoint): Mean of 9-point Self Measured Plasma Glucose Profile (SMPG) at Week 78
Description: Mean of the SMPG at 78 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime, at 4 am, before breakfast.
Time Frame: Week 78
Population: The FAS included all randomised subjects in the main trial including subjects carried through to the extension trial and missing data was imputed using LOCF. For 36 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 716 | 240
mmol/L | 7.2 (1.9) | 6.8 (1.4)

5. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 78 + 7 days follow up
Population: Safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or its comparator in the main trial including subjects carried through to the extension trial.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 753 | 251
Episodes/100 years of patient exposure | 1039 | 1271

6. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes are defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 78 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator in the main trial including subjects carried through to the extension trial.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 753 | 251
Episodes/100 years of patient exposure | 134 | 176

7. Primary Outcome: Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Mild AEs: no or transient symptoms, no interference with subject's daily activities. Moderate AEs: marked symptoms, moderate interference with subject's daily activities. Severe AEs: considerable interference with subject's daily activities, unacceptable. Serious adverse event (SAE): AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 78 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 753 | 251
Events/100 years of patient exposure
  Adverse events (AEs) | 411 | 403
  Serious AE | 20 | 20
  Severe AE | 24 | 20
  Moderate AE | 113 | 118
  Mild AE | 274 | 266
  Fatal AE | 1 | 1

8. Secondary Outcome: Main Trial (Secondary Endpoint): Rate of Confirmed Hypoglycaemic Episodes
Description: as for outcome 5
Time Frame: Week 0 to Week 52 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 753 | 251
Episodes/100 years of patient exposure | 1109 | 1363

9. Secondary Outcome: Main Trial (Secondary Endpoint): Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: as for outcome 6
Time Frame: Week 0 to Week 52 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 753 | 251
Episodes/100 years of patient exposure | 139 | 184

ADVERSE EVENTS:
Time Frame: Adverse events were collected in a time frame of 78 weeks + 7 days follow up.
Description: The SAS included all subjects who received at least one dose of investigational product or its comparator.
Arm/Group | IDeg OD | IGlar OD
Serious Adverse Events (participants affected / at risk) | 139/753 | 53/251
Other Adverse Events (participants affected / at risk) | 447/753 | 146/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=753) | IGlar OD (N=251)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (2)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (3) | 0 (0)
Angina unstable (Cardiac disorders) | 3 (3) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 8 (9) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 3 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0)
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (4) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Incision site abscess (Infections and infestations) | 1 (1) | 0 (0)
Infected sebaceous cyst (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Salmonella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 13 (13) | 2 (2)
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 6 (10) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Eating disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax spontaneous tension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adhesion (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) — Cause: Unknown
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Cholecystitis infective (Hepatobiliary disorders) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fibular fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
B cell lymphoma stage-1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastasis to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue carcinoma stage-1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Inter capillary glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Diastolic hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=753) | IGlar OD (N=251)
Diarrhoea (Gastrointestinal disorders) | 59 (73) | 26 (31)
Oedema peripheral (General disorders) | 55 (69) | 17 (20)
Influenza (Infections and infestations) | 58 (68) | 20 (23)
Nasopharyngitis (Infections and infestations) | 124 (212) | 37 (61)
Upper respiratory tract infection (Infections and infestations) | 123 (212) | 42 (70)
Wrong drug administered (Injury, poisoning and procedural complications) | 58 (66) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 (55) | 26 (36)
Back pain (Musculoskeletal and connective tissue disorders) | 56 (66) | 21 (25)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 47 (55) | 19 (19)
Headache (Nervous system disorders) | 71 (153) | 20 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 61 (71) | 21 (29)
Hypertension (Vascular disorders) | 50 (59) | 14 (15)
Vomiting (Gastrointestinal disorders) | 28 (39) | 14 (20)
Nausea (Gastrointestinal disorders) | 39 (45) | 15 (18)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 49 (64) | 13 (19)
Sinusitis (Infections and infestations) | 45 (64) | 18 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.